CLINICAL TRIAL: NCT01529125
Title: ART Pharmacokinetics, Mitochondrial Integrity, and Antioxidant Capacity in Severely Malnourished HIV-infected Malawian Children
Brief Title: Safety and Metabolic Study of Highly Active Antiretroviral Therapy (HAART) in Malnourished Children With HIV
Acronym: ARMAM
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ARTMAM
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Kwashiorkor; Marasmus; Severe Acute Malnutrition; HIV
MeSH Terms: conditions — Kwashiorkor; Protein-Energy Malnutrition; Severe Acute Malnutrition | interventions — Zidovudine; Lamivudine; Nevirapine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Kwashiorkor: HIV-positive children aged 6-59 months with kwashiorkor receiving nutritional rehabilitation and who are started on HAART.
  Interventions: Drug: zidovudine, lamivudine, nevirapine
- Marasmus: HIV-positive children aged 6-59 months with marasmus receiving nutritional rehabilitation and who are started on HAART.
  Interventions: Drug: zidovudine, lamivudine, nevirapine
- Control: HIV-positive children aged 6-59 months who are not severely malnourished and who are started on HAART for a non-nutritional reason.
  Interventions: Drug: zidovudine, lamivudine, nevirapine

INTERVENTIONS:
Drug: zidovudine, lamivudine, nevirapine

SUMMARY:
It is unclear whether children with HIV and severe acute malnutrition can be started on highly active antiretroviral therapy (HAART) safely while they are still malnourished and the manner in which this therapy should start. This study will examine the safety, efficacy, and metabolism of children started on HAART while still severely malnourished.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected about to start on HAART for the first time
* 6-59 months old

Exclusion Criteria:

* also being treated for TB
* other chronic illness (e.g., congenital heart disease, cerebral palsy)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6-59 months with HIV and kwashiorkor and marasmus who are not currently on HAART will be recruited from the Nutritional Rehabilitation Unit at Queen Elizabeth Central Hospital in Blantyre, Malawi. Controls will be recruited from the outpatient cotrimoxazole clinic who are about to start on HAART for a non-nutritional reason.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 6 weeks
  PK of ART in malnourished children

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi